CLINICAL TRIAL: NCT01765556
Title: A Phase I, Open-Label, Multicenter, Three-Period, One-Sequence Study To Investigate The Effect Of Ketoconazole On The Pharmacokinetics Of A Single Oral Dose Of 960 Mg Of Vemurafenib
Brief Title: A Pharmacokinetics Study to Investigate the Effect of Ketoconazole on Vemurafenib in Patients With BRAFV600 Mutation-Positive Metastatic Melanoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO28054; 2012-003143-29 (EudraCT Number)
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Malignant Melanoma, Neoplasms
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — Ketoconazole; Vemurafenib

ARMS (2):
- Ketoconazole treatment (Experimental)
  Interventions: Drug: ketoconazole
- Vemurafenib treatment (Experimental)
  Interventions: Drug: vemurafenib

INTERVENTIONS:
Drug: ketoconazole — multiple doses of ketoconazole in Period B and C
  Arms: Ketoconazole treatment
Drug: vemurafenib — single dose of vemurafenib in Period A and C
  Arms: Vemurafenib treatment

SUMMARY:
This open-label, multi-center, three-period, one sequence study will investigate the effect of ketoconazole on the pharmacokinetics of vemurafenib in patients with unresectable BRAFV600-mutation positive metastatic melanoma or other malignant tumor type that harbors a V600-activating mutation of BRAF without acceptable standard treatment options. Patients will receive a single dose of vemurafenib in Periods A and C and multiple doses of ketoconazole in Periods B and C. Eligible patients will have the option to continue treatment with vemurafenib as part of an extension study (NCT01739764). The anticipated time on study treatment is approximately 19 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >= 18 years old
* Patients with either unresectable Stage IIIc or Stage IV metastatic melanoma positive for the BRAFV600 mutation or other malignant tumor type that harbors a V600-activating mutation of BRAF, as determined by results of cobas® 4800 BRAF V600 mutation test or a DNA sequencing method, and who have no acceptable standard treatment options
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Life expectancy >= 12 weeks
* Full recovery from the effects of any major surgery or significant traumatic injury within 14 days prior to the first dose of study treatment
* Adequate hematologic and end organ function
* Female patients of childbearing potential and male patients with partners of childbearing potential must agree to always use two effective methods of contraception
* Negative serum pregnancy test within 7 days prior to commencement of dosing in women of childbearing potential

Exclusion Criteria:

* Prior treatment with vemurafenib or other BRAF inhibitor within 42 days of first dose of study drug
* Requirement for immediate or urgent treatment with daily vemurafenib and for whom the intermittent schedule of vemurafenib employed during the 19-day period for this trial is not clinically acceptable
* Allergy or hypersensitivity to components of the vemurafenib formulation
* Experimental therapy within 4 weeks prior to first dose of study drug
* Major surgical procedure or significant traumatic injury within 14 days prior to first dose of study drug or anticipation of the need for major surgery during study treatment
* Prior anti-cancer therapy within 28 days before the first dose of study drug
* History of clinically significant cardiac or pulmonary dysfunction
* History of symptomatic congestive heart failure of any New York Heart Association class or serious cardiac arrhythmia requiring treatment
* History of myocardial infarction within 6 months prior to first dose of study drug
* Current dyspnea at rest, owing to complications of advanced malignancy or any requirement for supplemental oxygen to perform activities of daily living
* History of congenital long QT syndrome or QTc > 450 ms
* Active central nervous system lesions
* Uncontrolled or poorly controlled diabetes
* Current severe, uncontrolled systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the concentration time curve | Approximately 19 days
Pharmacokinetics: Maximum plasma concentration | Approximately 19 days
Pharmacokinetics: Time to maximum plasma concentration | Approximately 19 days
Pharmacokinetics: Terminal half-life | Approximately 19 days
Pharmacokinetics: Apparent clearance | Approximately 19 days

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | Approximately 19 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche